CLINICAL TRIAL: NCT04493502
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of LY3041658 in Adults With Moderate-to-Severe Hidradenitis Suppurativa
Brief Title: A Study of LY3041658 in Adults With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17497; I7P-MC-DSAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-07-29; First posted 2020-07-30 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04-01

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3041658 (Experimental): Participants received 600 mg LY3041658 administered intravenously (IV) once every 2 weeks (Q2W).
  Interventions: Drug: LY3041658
- Placebo (Placebo Comparator): Placebo administered IV. Participants will switch to 600 mg LY3041658 administered IV after week 16.
  Interventions: Drug: Placebo; Drug: LY3041658

INTERVENTIONS:
Drug: Placebo — Administered IV
  Arms: Placebo
Drug: LY3041658 — Administered IV

SUMMARY:
The reason for this study is to see if the study drug LY3041658 is effective in participants with moderate-to-severe hidradenitis suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HS for at least 6 months
* Have HS lesions in at least 2 different anatomic areas
* Have inadequate response or intolerance to a 28 day course of oral antibiotics
* Have a total count of abscesses and inflammatory nodules greater than or equal to 4
* Agree to use a topical antiseptic daily
* Agree to stop using topical antibiotics during the study. In certain cases, oral antibiotics will be allowed

Exclusion Criteria:

* Have more than 20 draining fistulae
* Have received any biologic medication (adalimumab, etc.) for the treatment of HS
* Plan to use oral opioids for HS-related pain during the study
* Uncontrolled depression or suicidal thoughts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- United States (15):
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Skin Care Research, Inc, Hollywood, Florida
  - Nova Clinical Research, LLC, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Marietta Dermatology Clinical Research, Marietta, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Allcutis Research, Inc., Beverly, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - ALLCUTIS Research, Portsmouth, New Hampshire
  - Duke University Medical Center, Durham, North Carolina
  - UC Physicians Office Dermatology, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
- Australia (5):
  - Westmead Hospital, Northmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, QID
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Holdsworth House Medical Practice, Sydney

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3041658 in Adults With Hidradenitis Suppurativa — https://trials.lillytrialguide.com/en-US/trial/1U6Tipcu8f5y3goGhoMTA1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive either 600 milligram (mg) LY3041658, or placebo in the double blind period (16 weeks).
Groups:
- Placebo/600 mg LY3041658: Participants received placebo administered intravenously (IV) once every 2 weeks (Q2W) for 16 weeks in double blind period.
  Participants who previously assigned to placebo in double blind period received 600 mg LY3041658 administered IV Q2W until the last dosing visit in open-label period.
  Follow-up Period: Participants did not receive study drug during this period.
- 600 mg LY3041658 / 600 mg LY3041658: Participants received 600 mg LY3041658 administered IV Q2W in double blind and open-label period.
  Follow-up Period: Participants did not receive study drug during this period.
Period: Double Blind Treatment (Week 0 - 16)
Arm/Group | Placebo/600 mg LY3041658 | 600 mg LY3041658 / 600 mg LY3041658
Started | 24 | 48
Received at Least One Dose of Study Drug | 22 | 45
Completed | 14 | 38
Not Completed | 10 | 10
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 3 | 4
Not completed — Other, Relocation | 0 | 1
Not completed — Other, Protocol Deviation | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Randomized but Never Treated | 2 | 3
Period: Open-label Extension (Week 16 - 36)
Arm/Group | Placebo/600 mg LY3041658 | 600 mg LY3041658 / 600 mg LY3041658
Started | 14 | 38
Received at Least One Dose of Study Drug | 13 | 36
Completed | 10 | 29
Not Completed | 4 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 8
Period: Post-treatment Follow-up (10 Weeks)
Arm/Group | Placebo/600 mg LY3041658 | 600 mg LY3041658 / 600 mg LY3041658
Started | 10 | 29
Completed | 8 | 24
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo/600 mg LY3041658: Participants received placebo administered intravenously (IV) once every 2 weeks (Q2W) for 16 weeks in double blind period.
  Participants who previously assigned to placebo in double blind period received 600 mg LY3041658 administered IV Q2W until the last dosing visit in open-label period.
- 600 mg LY3041658 / 600 mg LY3041658: Participants received 600 mg LY3041658 administered IV Q2W in double blind and open-label period.
- Total: Total of all reporting groups
Arm/Group | Placebo/600 mg LY3041658 | 600 mg LY3041658 / 600 mg LY3041658 | Total
Number analyzed (Participants) | 22 | 45 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.10 (12.68) | 37.10 (12.38) | 36.80 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 35 | 47
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 15 | 35 | 50
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 12 | 17
  White | 16 | 30 | 46
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 2 | 5 | 7
  United States | 20 | 40 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 16
Description: The HiSCR is defined as at least a 50% reduction in the total abscess and inflammatory nodule count (sum of abscesses and inflammatory nodules [AN count]) with no increase in abscess count (A count) and no increase in draining fistulae count (DF count) relative to baseline. Non-responder imputation (NRI): Participants with missing data were considered non-responders.
Time Frame: Week 16
Population: Modified Intent-to-Treat (mITT) Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received placebo administered IV Q2W for 16 weeks.
- 600 mg LY3041658: Participants received 600 mg LY3041658 administered IV Q2W for 16 weeks.
Arm/Group | Placebo | 600 mg LY3041658
Number analyzed (Participants) | 22 | 45
percentage of participants | 31.8 [12.4 to 51.3] | 48.9 [34.3 to 63.5]
Statistical Analysis 1: Comparison: Placebo vs 600 mg LY3041658; Test type: Superiority; p = 0.189, Regression, Logistic; Mean Difference (Final Values) = 17.1, 95% CI 2-sided [-7.3 to 41.4]

2. Secondary Outcome: Mean Change From Baseline to Week 16 in Total Number of Abscesses and Inflammatory Nodules (AN) Count
Description: Mean Change from baseline in total AN count at Week 16 was reported. Abscess and inflammatory nodule were counted for the Hidradenitis Suppurativa (HS) affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Baseline, Week 16
Population: mITT Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: count of abscess and inflammatory nodule
Arm/Group | Placebo | 600 mg LY3041658
Number analyzed (Participants) | 22 | 45
count of abscess and inflammatory nodule | -1.85 (1.636) | -6.52 (1.133)
Statistical Analysis 1: Comparison: Placebo vs 600 mg LY3041658; Test type: Superiority; p = 0.024, ANCOVA; Mean Difference (Final Values) = -4.67, 95% CI 2-sided [-8.69 to -0.64]

3. Secondary Outcome: Mean Change From Baseline to Week 16 in Skin Pain on the HS Numeric Rating Scale (NRS)
Description: The Skin Pain - HS Numeric Rating Scale (NRS) is a patient-administered, single-question, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no skin pain" and 10 representing "skin pain as bad as you can imagine." The recall period is 7 days.
Time Frame: Baseline, Week 16
Population: mITT Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 600 mg LY3041658
Number analyzed (Participants) | 22 | 45
units on a scale | -1.83 (0.614) | -1.78 (0.418)
Statistical Analysis 1: Comparison: Placebo vs 600 mg LY3041658; Test type: Superiority; p = 0.949, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-1.44 to 1.53]

ADVERSE EVENTS:
Time Frame: Baseline Up to Follow-up Period (46 weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- 600 mg LY3041658 _Double-Blind Treatment Period: Participants received 600 mg LY3041658 IV Q2W for 16 weeks.
- Placebo_Double-Blind Treatment Period: Participants received placebo IV Q2W for 16 weeks.
- 600 mg LY3041658_Open-Label Extension: Participants received 600 mg IV LY3041658 Q2W from week 16-34 weeks.
- Follow-Up Period: Participants did not receive study drug during this period.
Arm/Group | 600 mg LY3041658 _Double-Blind Treatment Period | Placebo_Double-Blind Treatment Period | 600 mg LY3041658_Open-Label Extension | Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/22 | 0/49 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/45 | 2/22 | 1/49 | 0/39
Other Adverse Events (participants affected / at risk) | 10/45 | 2/22 | 13/49 | 2/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600 mg LY3041658 _Double-Blind Treatment Period (N=45) | Placebo_Double-Blind Treatment Period (N=22) | 600 mg LY3041658_Open-Label Extension (N=49) | Follow-Up Period (N=39)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 600 mg LY3041658 _Double-Blind Treatment Period (N=45) | Placebo_Double-Blind Treatment Period (N=22) | 600 mg LY3041658_Open-Label Extension (N=49) | Follow-Up Period (N=39)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1/10 (1) | 0/10 (0) | 0/12 (0) | 0/11 (0)
Scrotal operation (Surgical and medical procedures) | 0/10 (0) | 1/10 (1) | 0/12 (0) | 0/11 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT04493502/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT04493502/SAP_001.pdf